CLINICAL TRIAL: NCT05532605
Title: Effects of Mindfulness Based Therapy on Patients Perception of Illness and Depression in Cardiac Rehabilitation Phase-i
Brief Title: Effects of Mindfulness Based Therapy on Illness and Depression in Cardiac Rehab Phase-i
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sonia Ilyas
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Coronary Artery Stenosis
Keywords: depression; cardiac rehabilitation; patient perception of illness; MBSR; IPQ; HRQOL; Mindfulness
MeSH Terms: conditions — Coronary Stenosis; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac rehab phase I protocols (Active Comparator): will be treated with cardiac rehab phase I protocols
  Interventions: Other: cardiac rehabilitation phase I protocols
- Cardiac rehab phase I protocols + Mindfullness base therapy (Experimental): will be treated with cardiac rehab phase I protocols along with Mindfullness base therapy
  Interventions: Other: Cardiac rehab phase I protocols + Mindfullness base therapy

INTERVENTIONS:
Other: cardiac rehabilitation phase I protocols — cardiac rehab phase I protocols: ankel pumps, limbs ROMs, bed mobility. Do 5-10 minutes daily of breath awareness practice on your own.
  Arms: Cardiac rehab phase I protocols
Other: Cardiac rehab phase I protocols + Mindfullness base therapy — cardiac rehab phase I protocols: ankel pumps, limbs ROMs, bed mobility. Do 5-10 minutes daily of breath awareness practice on your own. Plus Mindfullness base therapy
  Arms: Cardiac rehab phase I protocols + Mindfullness base therapy

SUMMARY:
A randomize controlled trial will be conducted at Punjab institute of cardiology hospital Lahore, through convenience sampling technique on 48 patients which will be allocated through simple random sampling through sealed opaque enveloped into group A and Group B. Pretreatment values of patients' blood pressure, RR, HR, will be recorded. And patient's perception of illness through Illness Perception Questionnaire (IPQ), PHQ9 for depression assessment and HRQOL for quality of life will be assessed before and after treatment. Group A will be treated with basic Phase-I cardiac rehabilitation. And Group B will be treated with basic Phase-I cardiac rehabilitation along with Mindfulness based therapy. Treatment evaluation will be done after 8 weeks. Data will be analyzed using SPSS software version 25. After assessing normality of data by Shapiro-Wilk test, it will be decided either parametric or non-parametric test will be use within a group or between two groups.

DETAILED DESCRIPTION:
Cardiac rehabilitation is becoming more widely acknowledged as an important part of the overall treatment plan for individuals with cardiovascular disease. Cardiac rehabilitation programs aim to reduce the physiological and psychological impacts of heart disease.

Anxiety, depression, cardiovascular disease, and suicide are among poor health outcomes of stress, which is a global public health issue. Depression, a disorder with a significant psychological burden, has been linked to an increased risk of cardiovascular disease.

Although the exact nature of the links between depression and coronary heart disease (CHD) has yet to be determined, these links are increasingly being highlighted. The aim of the study is to find Effects of Mindfulness based therapy on patient perception of illness and depression in cardiac rehabilitation Phase-I.

A randomize controlled trial will be conducted at Punjab institute of cardiology hospital Lahore, through convenience sampling technique on 48 patients which will be allocated through simple random sampling through sealed opaque enveloped into group A and Group B. Pretreatment values of patients' blood pressure, RR, HR, will be recorded. And patient's perception of illness through Illness Perception Questionnaire (IPQ), PHQ9 for depression assessment and HRQOL for quality of life will be assessed before and after treatment. Group A will be treated with basic Phase-I cardiac rehabilitation. And Group B will be treated with basic Phase-I cardiac rehabilitation along with Mindfulness based therapy. Treatment evaluation will be done after 8 weeks. Data will be analyzed using SPSS software version 25. After assessing normality of data by Shapiro-Wilk test, it will be decided either parametric or non-parametric test will be use within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Phase-I CABG
* Hypertensive patients
* DM
* Patients hemodynamically stable

Exclusion Criteria:

* Hemodynamically unstable patients
* Orthopedic conditions i.e. fracture
* Disorientated patients
* Neuromuscular disease
* pacemaker dependency
* Uncontrolled arrhythmias
* Red Flags Like: Fever, Night Sweats, Malaise

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Illness perception questionnaire | 4 months
  The model proposes that situational stimuli (such as symptoms) generate both cognitive and emotional representations of the illness or health threat. These representations are processed in parallel through three stages. 0 is minimum and 10 is maximum.
PHQ9 for depression assessment | 4 months
  The Patient Health Questionnaire-9 (PHQ-9) is a nine-item questionnaire used in primary care and other medical settings to assess for depression. and The conventional cut-off score for detecting suspected major depression is 10 or higher. The Brief IPQ is a frequently used questionnaire with excellent psychometric qualities

SECONDARY OUTCOMES:
HRQOL for quality of life | 4 months
  Contemporary interpretations of HRQOL are based on the World Health Organization's definition of health as a state of complete physical, mental, and social well-being and not merely the absence of disease. contemporary HRQOL instrument domains are scored with a range of 0-100, with higher values representing better outcomes.
  To make useful inferences regarding absolute scores or change scores over time

CONTACTS AND LOCATIONS:
Overall Officials: Wajeeha Zia, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Punjab institute of cardiology hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wenger NK. Current status of cardiac rehabilitation. J Am Coll Cardiol. 2008 Apr 29;51(17):1619-31. doi: 10.1016/j.jacc.2008.01.030. PMID 18436113
- [Background] Dalal HM, Doherty P, Taylor RS. Cardiac rehabilitation. BMJ. 2015 Sep 29;351:h5000. doi: 10.1136/bmj.h5000. No abstract available. PMID 26419744
- [Background] Heran BS, Chen JM, Ebrahim S, Moxham T, Oldridge N, Rees K, Thompson DR, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2011 Jul 6;(7):CD001800. doi: 10.1002/14651858.CD001800.pub2. PMID 21735386
- [Background] Goel K, Pack QR, Lahr B, Greason KL, Lopez-Jimenez F, Squires RW, Zhang Z, Thomas RJ. Cardiac rehabilitation is associated with reduced long-term mortality in patients undergoing combined heart valve and CABG surgery. Eur J Prev Cardiol. 2015 Feb;22(2):159-68. doi: 10.1177/2047487313512219. Epub 2013 Nov 21. PMID 24265289
- [Background] Romas JA, Sharma M. Practical stress management: A comprehensive workbook: Academic Press; 2017.
- [Background] Milczarek M, González ER, Schneider E. OSH in figures: Stress at work-facts and figures: Office for Official Publ. of the Europ. Communities; 2009.
- [Background] Sharma M, Rush SE. Mindfulness-based stress reduction as a stress management intervention for healthy individuals: a systematic review. J Evid Based Complementary Altern Med. 2014 Oct;19(4):271-86. doi: 10.1177/2156587214543143. Epub 2014 Jul 22. PMID 25053754
- [Background] Nijjar PS, Connett JE, Lindquist R, Brown R, Burt M, Pergolski A, Wolfe A, Balaji P, Chandiramani N, Yu X, Kreitzer MJ, Everson-Rose SA. Randomized Trial of Mindfulness-Based Stress Reduction in Cardiac Patients Eligible for Cardiac Rehabilitation. Sci Rep. 2019 Dec 5;9(1):18415. doi: 10.1038/s41598-019-54932-2. PMID 31804580
- [Background] Rao A, Zecchin R, Newton PJ, Phillips JL, DiGiacomo M, Denniss AR, Hickman LD. The prevalence and impact of depression and anxiety in cardiac rehabilitation: A longitudinal cohort study. Eur J Prev Cardiol. 2020 Mar;27(5):478-489. doi: 10.1177/2047487319871716. Epub 2019 Oct 9. PMID 31597473
- [Background] Chauvet-Gelinier JC, Bonin B. Stress, anxiety and depression in heart disease patients: A major challenge for cardiac rehabilitation. Ann Phys Rehabil Med. 2017 Jan;60(1):6-12. doi: 10.1016/j.rehab.2016.09.002. Epub 2016 Oct 19. PMID 27771272
- [Background] Vieira A, Melo C, Machado J, Gabriel J. Virtual reality exercise on a home-based phase III cardiac rehabilitation program, effect on executive function, quality of life and depression, anxiety and stress: a randomized controlled trial. Disabil Rehabil Assist Technol. 2018 Feb;13(2):112-123. doi: 10.1080/17483107.2017.1297858. Epub 2017 Mar 13. PMID 28285574
- [Background] Kraal JJ, Van den Akker-Van Marle ME, Abu-Hanna A, Stut W, Peek N, Kemps HM. Clinical and cost-effectiveness of home-based cardiac rehabilitation compared to conventional, centre-based cardiac rehabilitation: Results of the FIT@Home study. Eur J Prev Cardiol. 2017 Aug;24(12):1260-1273. doi: 10.1177/2047487317710803. Epub 2017 May 23. PMID 28534417
- [Background] Kachur S, Menezes AR, De Schutter A, Milani RV, Lavie CJ. Significance of Comorbid Psychological Stress and Depression on Outcomes After Cardiac Rehabilitation. Am J Med. 2016 Dec;129(12):1316-1321. doi: 10.1016/j.amjmed.2016.07.006. Epub 2016 Jul 30. PMID 27480388
- [Background] Blumenthal JA, Sherwood A, Smith PJ, Watkins L, Mabe S, Kraus WE, Ingle K, Miller P, Hinderliter A. Enhancing Cardiac Rehabilitation With Stress Management Training: A Randomized, Clinical Efficacy Trial. Circulation. 2016 Apr 5;133(14):1341-50. doi: 10.1161/CIRCULATIONAHA.115.018926. Epub 2016 Mar 21. PMID 27045127
- [Background] Shields GE, Wells A, Doherty P, Heagerty A, Buck D, Davies LM. Cost-effectiveness of cardiac rehabilitation: a systematic review. Heart. 2018 Sep;104(17):1403-1410. doi: 10.1136/heartjnl-2017-312809. Epub 2018 Apr 13. PMID 29654096
- [Background] Broadbent E, Wilkes C, Koschwanez H, Weinman J, Norton S, Petrie KJ. A systematic review and meta-analysis of the Brief Illness Perception Questionnaire. Psychol Health. 2015;30(11):1361-85. doi: 10.1080/08870446.2015.1070851. Epub 2015 Aug 26. PMID 26181764
- [Background] Knapen J, Vancampfort D, Morien Y, Marchal Y. Exercise therapy improves both mental and physical health in patients with major depression. Disabil Rehabil. 2015;37(16):1490-5. doi: 10.3109/09638288.2014.972579. Epub 2014 Oct 24. PMID 25342564
- [Background] Jolly K, Lip GY, Sandercock J, Greenfield SM, Raftery JP, Mant J, Taylor R, Lane D, Lee KW, Stevens AJ. Home-based versus hospital-based cardiac rehabilitation after myocardial infarction or revascularisation: design and rationale of the Birmingham Rehabilitation Uptake Maximisation Study (BRUM): a randomised controlled trial [ISRCTN72884263]. BMC Cardiovasc Disord. 2003 Sep 10;3:10. doi: 10.1186/1471-2261-3-10. Epub 2003 Sep 10. PMID 12964946
- [Background] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240
- [Background] Martin A, Rief W, Klaiberg A, Braehler E. Validity of the Brief Patient Health Questionnaire Mood Scale (PHQ-9) in the general population. Gen Hosp Psychiatry. 2006 Jan-Feb;28(1):71-7. doi: 10.1016/j.genhosppsych.2005.07.003. PMID 16377369
- [Background] Moriarty DG, Zack MM, Kobau R. The Centers for Disease Control and Prevention's Healthy Days Measures - population tracking of perceived physical and mental health over time. Health Qual Life Outcomes. 2003 Sep 2;1:37. doi: 10.1186/1477-7525-1-37. PMID 14498988
- [Background] Bishop SR. What do we really know about mindfulness-based stress reduction? Psychosom Med. 2002 Jan-Feb;64(1):71-83. doi: 10.1097/00006842-200201000-00010. PMID 11818588